CLINICAL TRIAL: NCT05344261
Title: Prophylactic Treatment of Neuroma and Phantom Limb Pain With Targeted Muscle Reinnervation (TMR) and Regenerative Peripheral Interface (RPNI) at the Time of Major Limb Amputation: A Randomized Control Trial
Brief Title: Effect of Prophylactic TMR and RPNI on Neuroma and Phantom Limb Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never initiated and no participants enrolled
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Travis Boyd, ASSISTANT PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2021-0348
Record Dates: First submitted 2022-03-28; First posted 2022-04-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Amputation; Neuroma Amputation; Phantom Limb Pain; Residual Limbs
Keywords: Targeted Muscle Re-innervation; Regenerative Peripheral Nerve Interface; TMR; RPNI
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Active Comparator): Standard Post-Amputation Surgical Care: Briefly, the transected nerves will be blindly tucked into surrounding bulky soft tissue to protect the nerve ends before the wound is closed.
  Interventions: Procedure: Standard Post-Amputation Surgical Care
- Targeted Muscle Re-innervation (Experimental): Briefly, each transected nerve is identified after amputation using 6-0 Prolene suture and is dissected proximally for length. With minimal dissection, a nerve stimulator is used to identify functional motor nerve branches. Near the point where the motor branch enters the muscle, the motor nerve branch is transected and an end-to-end coaptation is performed with a nearby tagged amputated nerve.
  Interventions: Procedure: Targeted Muscle Re-innervation
- Regenerative Peripheral Nerve Interface (Experimental): Briefly, a muscle graft (usually from the amputated limb) is wrapped around the clean ends of the transected nerve(s).
  Interventions: Procedure: Regenerative Peripheral Nerve Interface

INTERVENTIONS:
Procedure: Targeted Muscle Re-innervation — Targeted Muscle Re-innervation involves re-routing transected nerve ends to functional motor nerves proximal to the site of amputation.
  Arms: Targeted Muscle Re-innervation
Procedure: Regenerative Peripheral Nerve Interface — Regenerative Peripheral Nerve Interface involves placing transected nerve ends in harvested muscle grafts.
  Arms: Regenerative Peripheral Nerve Interface
Procedure: Standard Post-Amputation Surgical Care — Standard post-amputation surgical care involves placing transected nerve ends into muscle/soft tissue proximal to the site of amputation.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to analyze the efficacy of novel interventions in post-amputation surgical care (specifically Targeted Muscle Reinnervation and Regenerative Peripheral Nerve Interface) on post-amputation pain and functional outcomes at the time of amputation. These novel interventions have been shown to be successful in treating the downstream effects of amputations (pain, phantom limb pain, neuroma pain, etc.), but has not been studied in a randomized manner at the time of amputation.

DETAILED DESCRIPTION:
The investigators plan a randomized control trial of all eligible patients undergoing major limb amputation at Parkland Memorial Hospital. Eligible patients undergoing an amputation will be consented for all possible interventions and randomized to either receive Targeted Muscle Re-Innervation (TMR), Regenerative Peripheral Nerve Interface (RPNI), or standard post-amputation surgical care at the time of their operation. Key pre-operative data including patient sex, age, BMI, past medical history, past surgical history, medications, allergies, social history, social support systems, exposure to narcotic medication, and reason for amputation will be analyzed. Intra-operatively, patients randomized to the treatment arm will receive TMR or RPNI and the transected nerve ends addressed will be recorded. Post-operative data that will be recorded include hospital stay, complications related to the procedure, complications leading to reoperation, functional results, need for pain medication, incidence of phantom limb pain, incidence of painful neuromas, length of follow-up, and all adverse events/complications. Analyses will be conducted using data obtained from patient medical records from the Parkland Health & Hospital System.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Patients scheduled for amputation of upper or lower extremity (including digit, ray, and hand) as a primary or secondary sequela of trauma.
* Patients scheduled for amputation of upper or lower extremity (including digit, ray, and hand) for primary or secondary sequelae of malignancy.
* Secondary sequalae include but is not limited to metastatic disease and osteolytic disease.
* Patients scheduled for amputation of upper or lower extremity (including digit, ray, and hand) for vasculitic diseases.

Exclusion Criteria:

* Patients less than 18 years old
* Patients with cognitive impairment
* Patients who are imprisoned at the time of randomization
* Patients currently enrolled in other studies relating to neuropathic pain
* Patients actively undergoing radiation therapy
* Patients with existing neuroma or underwent prior neuroma surgery
* Patients with amputations scheduled congenital reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Phantom Limb Pain | Specifically at the time point 1 year after their primary incisions have healed.
  The primary outcome measure of the study will the incidence of phantom limb pain in each group over the course of the recovery period.

SECONDARY OUTCOMES:
Pain intensity score as measured PROMIS (Patient Reported Outcomes Measurement Information System) score | Until 2 years after incisions have healed.
  Pain intensity score is measured bv PROMIS (Patient Reported Outcomes Measurement Information System) Scores via patient questionnaires administered at follow-up visits. Possible scores range from 1-5 where higher scores indicate worse outcome (pain severity).
Pain interference score as measured by PROMIS (Patient Reported Outcomes Measurement information System) questionnaire | Until 2 years after incisions have healed.
  Pain interference score as measured by PROMIS (Patient Reported Outcomes Measurement information System) scores via patient questionnaires administered at follow-up visits. Possible scores range from 1-5, where higher scores indicate worse outcome (pain interference).
Pain behavior measured by PROMIS (Patient Reported Outcomes Measurement Information System) questionnaire | Until 2 years after incisions have healed.
  Pain behavior score measured by PROMIS (Patient Reported Outcomes Measurement Information System) questionnaire that pertains to subject social health. Raw summed score from 8 to 40, where 40 represents severely maladaptive pain behavior.
Narcotic medical use post-operatively as measured by MME (Morphine Milligram Equivalent) Score | Until 2 years after incisions have healed.
  Narcotic medical use post-operatively as measured by MME (Morphine Milligram Equivalent) Score This is a tool to condense and standardize the patient's narcotic pain regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Noble, Study Director — UT Southwestern Department of Plastic Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Dumanian GA, Potter BK, Mioton LM, Ko JH, Cheesborough JE, Souza JM, Ertl WJ, Tintle SM, Nanos GP, Valerio IL, Kuiken TA, Apkarian AV, Porter K, Jordan SW. Targeted Muscle Reinnervation Treats Neuroma and Phantom Pain in Major Limb Amputees: A Randomized Clinical Trial. Ann Surg. 2019 Aug;270(2):238-246. doi: 10.1097/SLA.0000000000003088. PMID 30371518
- [Background] Valerio IL, Dumanian GA, Jordan SW, Mioton LM, Bowen JB, West JM, Porter K, Ko JH, Souza JM, Potter BK. Preemptive Treatment of Phantom and Residual Limb Pain with Targeted Muscle Reinnervation at the Time of Major Limb Amputation. J Am Coll Surg. 2019 Mar;228(3):217-226. doi: 10.1016/j.jamcollsurg.2018.12.015. Epub 2019 Jan 8. PMID 30634038
- [Background] Eberlin KR, Ducic I. Surgical Algorithm for Neuroma Management: A Changing Treatment Paradigm. Plast Reconstr Surg Glob Open. 2018 Oct 16;6(10):e1952. doi: 10.1097/GOX.0000000000001952. eCollection 2018 Oct. PMID 30534497
- [Background] Kubiak CA, Kemp SWP, Cederna PS, Kung TA. Prophylactic Regenerative Peripheral Nerve Interfaces to Prevent Postamputation Pain. Plast Reconstr Surg. 2019 Sep;144(3):421e-430e. doi: 10.1097/PRS.0000000000005922. PMID 31461024
- [Background] Santosa KB, Oliver JD, Cederna PS, Kung TA. Regenerative Peripheral Nerve Interfaces for Prevention and Management of Neuromas. Clin Plast Surg. 2020 Apr;47(2):311-321. doi: 10.1016/j.cps.2020.01.004. Epub 2020 Feb 1. PMID 32115057
- [Background] Kuiken TA, Barlow AK, Hargrove L, Dumanian GA. Targeted Muscle Reinnervation for the Upper and Lower Extremity. Tech Orthop. 2017 Jun;32(2):109-116. doi: 10.1097/BTO.0000000000000194. PMID 28579692